CLINICAL TRIAL: NCT04628455
Title: Needlescopic Inversion and Snaring for Inguinal Hernia in Girls Using 1.6-mm Instruments
Brief Title: Needlescopic Inversion and Snaring of Hernia in Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Rafik Shalaby, Professor of Pediatric Surgery, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS2020-1002
Record Dates: First submitted 2020-05-15; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Inguinal Hernia; Polyps; Fallopian Tube Injury; Round Ligament; Anomaly
MeSH Terms: conditions — Hernia, Inguinal; Polyps; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Both SGDs were used to invert the hernia sac by gradual sustained alternating traction on the round ligament. Each SGD hands to the other one till complete inversion occurs, this is known by the hernial sac hanging from internal ring without retracting-back inside the inguinal canal. . SGD-C passed inside the loop of MPS and re-catches the hernial sac, which is then twisted around its neck several times. MPS is closed tightly at the proper neck and coagulation diathermy current is applied.Detached sac was then pushed antigradely out through the umbilical port.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inversion and Snaring (Other): needlescopic inversion, snaring, and excision of the hernia sac using two Suture Grasper Sevice of Mediflex Company and a home made snare
  Interventions: Device: Inversion and snaring

INTERVENTIONS:
Device: Inversion and snaring — Vertical umbilical 5-mm incision was made for 5-mm trocar. Pneumoperitoneum is then established with CO2 flow of 1.5-2.5 L/min keeping intraabdominal pressure between 8-12 mmHg. A two-mm incision was done at a point B [midway between umbilicus and symphysis pubis] for 2-mm port passed under direct vision and a tiny 11-blade scalpel puncture is done at the corresponding Mac-Burney's [Point C] for SGD.
  Both SGDs were used to invert the hernia sac by gradual sustained alternating traction on the round ligament. Each SGD hands to the other one till complete inversion occurs, this is known by the hernial sac hanging from internal ring without retracting-back inside the inguinal canal. Then, the MPS is introduced via 2-mm trocar at point. SGD-C passed inside the loop of MPS and re-catches the hernial sac, which is then twisted around its neck several times. MPS was closed at the neck and diathermy current is applied. Detached sac was then pushed antigradely out through the umbilical port.

SUMMARY:
Two Millimetres needlescopic instruments induce minimal damage to the abdominal wall and have excellent cosmetic results. However, these instruments are fragile and expensive with short weak jaws. The aim of this study is to present a novel needlescopic approach using 1.6-mm Suture Grasper Device [SGD], modified polypectomy snare and a home-made Snare (HMS) for the treatment of congenital inguinal hernias [CIH] in girls. Over a period of one year from March 2018 to March 2019 a prospective study was conducted in three tertiary centres on 53 girls presented with CIH. Preoperative inguinoscrotal U/S was done for all patients to confirm the diagnosis and to measure the diameter of internal inguinal ring [IIR]. All patients were repaired using needlescopic inversion and snaring of the hernia sac using 2-SGDs and a snare. Follow up period ranged from 12 to 24 (Median 16.5) months. Fifty-three girls with 74 hernias were included in this study. Their mean age was 37.8 months. Internal inguinal ring diameter (IIR) ranged between 8-15 mm with a mean of 11.8±2.8mm. Mean operative time was 15.5 minutes in bilateral and 11.4 minutes in unilateral cases. Mean operative time for inversion, snaring, and sac extraction was 4.2±1.3 minutes. All cases were completed successfully without conversion and without complications. Follow up period ranged from 12 to 24 (Median 16.5) months with non-visible scar and no recurrence among the studied patients. Needlescopic inversion and snaring of inguinal hernia using 1.6mm instruments is a safe, rapid and feasible method for CIH repair in girls with invisible scar and no short-term recurrence.

DETAILED DESCRIPTION:
Operative details: Patient lies in supine position at upper part of OR table towards right edge. Operating table is tilted to opposite side of hernia with 30-degree Trendelenburg position. Operator stands on patient's right side during either uni-or bi-lateral hernia. Camera man stands at table head and monitor facing patient's feet. Vertical trans umbilical 5-mm incision [Point A] was made and 5-mm trocar passed under vision using open technique. Pneumoperitoneum is then established with CO2 flow of 1.5-2.5 L/min keeping intraabdominal pressure between 8-12 mmHg according to patients' age and weight. Early in our experience, a two-mm incision is done at a point located midway between umbilicus and symphysis pubis [point B] for 2-mm port passed under direct vision and a tiny 11-blade scalpel puncture was done at the corresponding Mac-Burney's [Point C] for SGD. Abdomen was then explored to confirm the diagnosis and detect contralateral or other hernias if present.

One SGD was introduced through point B (SGD-B) and another one through point C (SGD-C). Both SGDs were used to invert the hernia sac by gradual sustained alternating traction on the round ligament. Each SGD hands to the other one till complete inversion occurs, this is known by the hernial sac hanging from internal ring without retracting-back inside the inguinal canal. Occasionally, investigators had to fix the sac to the anterior abdominal wall by a suture [Prolne 2/0 on a half circle 20-mm needle] placed percutaneously lateral to the corresponding Mac-Berney's point to prevent its retraction. Then, the MPS was introduced via the trocar at point B and opened inside the abdomen and SGD-C passed inside the loop of MPS and re-catches the hernial sac, which is then twisted around its neck several times. MPS was closed tightly at the proper neck and coagulation diathermy current is applied to it leading to separation of the hernia sac. Detached sac (grasped by SGD-C) was then pushed antegradely out through the umbilical port. In some cases, the Fallopian's tube was closely related to the round ligament and investigators had to divide the round ligament with the long microdiathermy needle introduced directly via point B before hernia sac snaring to avoid its injury during the application of MPS. Deflation of the abdomen is done, and umbilical fascial incision is closed using 2/0 or 3/0 Polygalctin suture and umbilical skin layers were closed using 4/0 Polygalctin suture. Later in the study, we were able to innovate a HMS by using the guide wire of central venous catheter looped through VAC and connected to a regular diathermy probe and investigators modified our technique. An11-blade scalpel puncture is done at point-B through which VAC is introduced directly instead of 2-mm trocar. This VAC is used for the insertion of HMS and SGD-B. Then, complete inversion of the sac was done using 2 SGDs as previously described. Followed by introduction of HMS through #14-G VAC at point-B and the procedure completed as before.

Postoperative Management:

Patients received antibiotics and analgesics according to hospital protocols. Oral fluids started 2 hours post operatively and diet was advanced gradually as tolerated. Patients were discharged the same post-operative day. Follow up period ranged from 12 to 24 (Median 16.5) months. with for recurrence and cosmetic results.

Discussion:

In the last 2 decades, pediatric inguinal hernia repair witnessed a huge evolution with laparoscopic approaches attracting more and more pediatric surgeons and laparoscopic hernia repair became well-established and popular technique with comparable recurrence rates and operative time. Moreover, laparoscopy allows diagnosis of contralateral and other coexisting hernia with a chance for simultaneous repair. Early in the laparoscopic era, its drawbacks were long learning curve, need for smaller instruments for younger kids, higher recurrence rates, and to somewhat smaller but visible scars compared to conventional open hernia repair. With time, regular use of laparoscopy, fine instruments, introduction of newer concepts and techniques for tailoring which laparoscopic technique fits for each patient the results came to be similar or even better than that of conventional repair. Laparoscopy for female inguinal hernia repair was first introduced in 1997 by El Gohary. He described hernial sac inversion and ligation in girls using 5-mm instruments and endo loop with excellent results.

During the evolution of laparoscopic repair of hernia, results improved very much by cautery of the IIR enhancing peritoneal fibrosis hence reducing recurrence rates compared to simple peritoneal closure.

Snaring is routinely used for colonic polypectomy with excision of polyps at its proper neck using coagulation current without colonic wall perforation. In this study it is proposed that inversion and snaring of the hernia sac results in a herniotomy with narrow raw area at its neck of the hernia sac combining the benefits of both peritoneal disconnection and thermal injury to prevent recurrence. Recently there is a report of early results of inversion, and snaring of hernial sac using 3-mm instruments and commercial polypectomy snare in girls with encouraging results and no recurrence. On application of monopolar diathermy current to the snare itself, the hernial sac will shrink with almost closure of internal ring. No recurrence was reported with no perioperative complications except for lymphocele developed at the level of labium major 2 weeks postoperatively that completely resolved after 6 months.

Commercially available polypectomy snare length is 230-cm which imposed discomfort and difficulty using it for hernial sac snaring. So, investigators opted to shorten it from 230-cm to 50 cm to facilitate its usage. The biomedical engineering department was contacted and succeeded to shorten it to the required length. In this study, in the first 2 months investigator used this modified snare successfully but it is still not fully satisfied as it adds extra cost [needs 2-mm trocar for insertion], needs technical assistance for shortening and re-sterilization. Investigator came into another innovation by developing a home-made snare (HMS) made of central venous catheter guide wire looped through VAC and connected to a regular diathermy probe. Each wire can be cut to make 2-3 snares. It is shorter, easy to use, cheaper and avoided the use of expensive trocar 2-mm. This HMS was then applied for all upcoming cases after that. It is well known that, one of the most annoying factors lead to delayed acceptance of laparoscopic repair for CIH among pediatric surgeons is visible scars even though they are smaller compared to the hidden skin crease scar of the open repair which ultimately resulted in development of needlescopic repair. Chock et al. reported that despite good cosmetic results, 2-mm instruments are expensive, delicate, flexible, and with short and weak jaws limiting their use on a wide scale. Others reported that needlescopic instruments can be used only by expert surgeons as it can be bended easily and its small jaws limit the power of grasping the tissue with unsuitability for ideal retraction and tissue handling. In contrary, SGD used for port closure is only 1.6 mm in diameter with adequate length, strong shaft, ergonomic handle, cheap, wide jaw and offers a very good tissue grip. According to the results of this study, needlescopic inversion, snaring and complete excision of the hernia is a progress of minilaparoscopic surgery where two MSDs [1.6-mm diameter] were used instead of 2-3-mm instruments for the treatment of CIH in girls. It avoids the disadvantages of 2-mm instruments.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral congenital inguinal hernia Unilateral congenital inguinal hernia Hernia defect siameter less than 1.5 mm

Exclusion Criteria:

* Recurrent hernia age less than 6 Month Contraindication to laparoscopy

Ages: 6 Months to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Bilateral inguinal hernia, Unilateral inguinal hernia
Enrollment: 53 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Recurrence of Hernia | every month up to one year postoperative
  All patients were examined clinical and by U/S for detection of the recurrence

SECONDARY OUTCOMES:
Operative time | every minute up to 2 hours (the end of the surgery)
  The operative time will be measured by minutes from the start of skin incision to the end of operation

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Y Shalaby, MD, Principal Investigator — Al-Azhar University
Locations (2):
- Egypt (2):
  - Rafik Sahalaby, Cairo
  - Rafik Shalaby, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McClain L, Streck C, Lesher A, Cina R, Hebra A. Laparoscopic needle-assisted inguinal hernia repair in 495 children. Surg Endosc. 2015 Apr;29(4):781-6. doi: 10.1007/s00464-014-3739-8. Epub 2014 Aug 9. PMID 25106720
- [Background] Schier F. Laparoscopic herniorrhaphy in girls. J Pediatr Surg. 1998 Oct;33(10):1495-7. doi: 10.1016/s0022-3468(98)90483-3. PMID 9802799
- [Result] Wang K, Cai J, Lu YC, Li XW, Zhai GM, He WB, Guo XS, Wu GQ. A Faster and Simpler Operation Method for Laparoscopic Inguinal Hernia Repair in Children. J Laparoendosc Adv Surg Tech A. 2020 Jun;30(6):706-711. doi: 10.1089/lap.2019.0598. Epub 2020 Mar 27. PMID 32216722
- [Result] Kantor N, Travis N, Wayne C, Nasr A. Laparoscopic versus open inguinal hernia repair in children: which is the true gold-standard? A systematic review and meta-analysis. Pediatr Surg Int. 2019 Sep;35(9):1013-1026. doi: 10.1007/s00383-019-04521-1. Epub 2019 Jul 10. PMID 31292721
- [Result] Chan IH, Tam PK. Laparoscopic Inguinal Hernia Repair in Infants and Children: State-of-the-Art Technique. Eur J Pediatr Surg. 2017 Dec;27(6):465-471. doi: 10.1055/s-0037-1608685. Epub 2017 Nov 22. No abstract available. PMID 29166678
- [Result] Gause CD, Casamassima MGS, Yang J, Hsiung G, Rhee D, Salazar JH, Papandria D, Pryor HI 2nd, Stewart D, Lukish J, Colombani P, Chandler NM, Johnson E, Abdullah F. Laparoscopic versus open inguinal hernia repair in children </=3: a randomized controlled trial. Pediatr Surg Int. 2017 Mar;33(3):367-376. doi: 10.1007/s00383-016-4029-4. Epub 2016 Dec 26. PMID 28025693
- [Result] Barroso C, Etlinger P, Alves AL, Osorio A, Carvalho JL, Lamas-Pinheiro R, Correia-Pinto J. Learning Curves for Laparoscopic Repair of Inguinal Hernia and Communicating Hydrocele in Children. Front Pediatr. 2017 Sep 27;5:207. doi: 10.3389/fped.2017.00207. eCollection 2017. PMID 29021976
- [Result] Zallen G, Glick PL. Laparoscopic inversion and ligation inguinal hernia repair in girls. J Laparoendosc Adv Surg Tech A. 2007 Feb;17(1):143-5. doi: 10.1089/lap.2006.0553. PMID 17362194
- [Result] Guner YS, Emami CN, Chokshi NK, Wang K, Shin CE. Inversion herniotomy: a laparoscopic technique for female inguinal hernia repair. J Laparoendosc Adv Surg Tech A. 2010 Jun;20(5):481-4. doi: 10.1089/lap.2009.0169. PMID 20367121
- [Result] Xi HW, Duan WQ, Cui QQ, You ZH, Zhao Z, Zhang P. Transumbilical Single-Site Laparoscopic Inguinal Hernia Inversion and Ligation in Girls. J Laparoendosc Adv Surg Tech A. 2015 Jun;25(6):522-5. doi: 10.1089/lap.2014.0383. Epub 2015 May 5. PMID 25941750
- [Result] Ostlie DJ, Ponsky TA. Technical options of the laparoscopic pediatric inguinal hernia repair. J Laparoendosc Adv Surg Tech A. 2014 Mar;24(3):194-8. doi: 10.1089/lap.2014.0081. PMID 24625350
- [Result] Lipskar AM, Soffer SZ, Glick RD, Rosen NG, Levitt MA, Hong AR. Laparoscopic inguinal hernia inversion and ligation in female children: a review of 173 consecutive cases at a single institution. J Pediatr Surg. 2010 Jun;45(6):1370-4. doi: 10.1016/j.jpedsurg.2010.02.113. PMID 20620347
- [Result] Chen YN, Chang LC, Chang CY, Chen PJ, Chen CY, Tseng CH, Chiu HM. Comparison of cold and hot snaring polypectomy for small colorectal polyps: study protocol for a randomized controlled trial. Trials. 2018 Jul 6;19(1):361. doi: 10.1186/s13063-018-2743-z. PMID 29980220
- [Result] Blatnik JA, Harth KC, Krpata DM, Kelly KB, Schomisch SJ, Ponsky TA. Stitch versus scar--evaluation of laparoscopic pediatric inguinal hernia repair: a pilot study in a rabbit model. J Laparoendosc Adv Surg Tech A. 2012 Oct;22(8):848-51. doi: 10.1089/lap.2012.0137. Epub 2012 Sep 18. PMID 22989037
- [Result] Shalaby R, Elsaied A, Shehata S, Shehata S, Hamed A, Alsamahy O, Ashour Y, Elsayaad I, Shahin M. Needlescopic assisted internal ring suturing; a novel application of low-cost home-made instruments for pediatric inguinal hernia repair. Hernia. 2019 Dec;23(6):1279-1289. doi: 10.1007/s10029-019-01982-0. Epub 2019 May 25. PMID 31129795
- [Result] Novotny NM, Puentes MC, Leopold R, Ortega M, Godoy-Lenz J. The Burnia: Laparoscopic Sutureless Inguinal Hernia Repair in Girls. J Laparoendosc Adv Surg Tech A. 2017 Apr;27(4):430-433. doi: 10.1089/lap.2016.0234. Epub 2017 Mar 30. PMID 28358588
- [Result] St-Louis E, Chabot A, Stagg H, Baird R. Experience with peritoneal thermal injury during subcutaneous endoscopically assisted ligation for pediatric inguinal hernia. J Pediatr Surg. 2018 May;53(5):968-972. doi: 10.1016/j.jpedsurg.2018.02.024. Epub 2018 Feb 9. PMID 29501237
- [Result] Chock A, Seslar S, Stoopen E, Tristan A, Hashish H, Gonzalez JJ, Franklin ME Jr. Needlescopic appendectomy. Surg Endosc. 2003 Sep;17(9):1451-3. doi: 10.1007/s00464-002-8732-y. Epub 2003 Jun 19. PMID 12811662
- [Result] Wada H, Kimura T, Kawabe A, Sato M, Miyaki Y, Tochikubo J, Inamori K, Shiiya N. Laparoscopic transabdominal preperitoneal inguinal hernia repair using needlescopic instruments: a 15-year, single-center experience in 317 patients. Surg Endosc. 2012 Jul;26(7):1898-902. doi: 10.1007/s00464-011-2122-2. Epub 2012 Jan 6. PMID 22223115
- [Result] Schier F. Laparoscopic appendectomy with 1.7-mm instruments. Pediatr Surg Int. 1998 Nov;14(1-2):142-3. doi: 10.1007/s003830050465. PMID 9880727
- [Result] Shalaby R, Abdalrazek M, Hamed A, Elhady S, Ibrahim R, Shahin M, Helal A, Elsaied A, Mohamad S, Mahfouz M, Elsherbeny M, El-Lithy MM. Novel application of the sewing machine principle; a new simplified intracorporeal suturing technique for pediatric inguinal hernia. J Pediatr Surg. 2019 Jul;54(7):1505-1509. doi: 10.1016/j.jpedsurg.2019.01.054. Epub 2019 Feb 18. PMID 30827487